CLINICAL TRIAL: NCT07051863
Title: Prospective Cohort and Biobank of Patients With Nonalcoholic Fatty Liver Disease (NAFLD Cohort Study)
Brief Title: Prospective Cohort and Biobank of Patients With Nonalcoholic Fatty Liver Disease
Acronym: NAFLD Cohort
Status: Recruiting | Type: Observational
Sponsor: Fondazione Epatocentro Ticino (Other)
Responsible Party: Sponsor
Other Study IDs: NAFLD Cohort Study
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: NAFLD; MASH; NASH/MASH
Keywords: NAFLD; MASH; NASH; Steatoepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Serum, whole blood sample, citrate sample, Paxgene blood RNA, fecal samples, urine samples, fragments of liver biopsy specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to establish a unified cohort for retrospective and prospective high quality baseline and follow-up data registration of patients with a diagnosis of NAFLD/NASH/MAFLD, according to standardized criteria.

This will allow future studies aimed at elucidate clinical presentation, natural history, response to treatment, genetic and metabolic risk factors, treatment options and outcomes of the disease. The cohort will allow investigators to carry out genetic, serological, microbiologic and immunological studies.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years of age at the time of signing the informed consent
2. Participant willing to sign the informed consent form (ICF) and to complete all study-specific procedures and visits
3. To have a diagnosis of NAFLD/NASH/MAFLD followed at Epatocentro Ticino and collaborating/referring clinicians based on:

   1. Liver biopsy with a histological evidence of NAFLD/NASH/MAFLD OR
   2. Liver imaging (ultrasound, CT scan, MRI, CAP Controlled Attenuation Parameter) OR
   3. Diagnosis of metabolic syndrome and liver fibrosis or cirrhosis without an alternative diagnosis; metabolic syndrome fulfilling one or more of the below mentioned conditions:

      * Abdominal obesity: a waist circumference of more than 35 inches (>89cm) for women and more than 40 inches (>102 cm) for men;
      * High blood pressure of 130/80 mm Hg or higher. Normal blood pressure is defined as less than 130 mm Hg for systolic pressure, and less than 80 mm Hg for diastolic pressure
      * Impaired fasting blood glucose. This means a level equal to or greater than 100 mg/dL (>5.6 mmol/L)
      * High triglyceride levels of more than 150 mg/dL (> 1.7mmol/L).
      * Low HDL (good) cholesterol: less than 40 mg/dL (< 1.04 mmol/L) for men and less than 50 mg/dL (< 1.29 mmol/L) for women
4. alcohol consumption less than 21 (males) or 14 (women) units per week in the 6 months before the enrolment and no history of excessive alcohol consumption in the 5 years before enrolment. One unit is 12g (grams) of pure alcohol; 10-12 grams of pure alcohol are contained in a 280-330 ml of beer, 150-180 ml of champagne, 30-40 ml of whisky or high-strength spirit, 60-80 ml of liqueur, and 100-120 ml of red wine

Exclusion Criteria:

1. To have a diagnosis of type I diabetes mellitus
2. To have a concomitant liver disease
3. To take or have taken in the last 12 months before enrolment, on more than 50% of days, drugs that may cause liver steatosis (long-term high dose systemic corticosteroids (> 20mg prednisone equivalent), amiodarone, methotrexate, tamoxifen, tetracycline, high dose estrogens and valproic acid)
4. Pregnancy and breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient wiht diagnosis of NAFLD/NASH/MAFLD
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Establish a unified cohort for retrospective and prospective data of patients with a diagnosis of NAFLD/NASH/MAFLD | 7 years
  The primary objective of this project is to establish a unified cohort for retrospective and prospective highquality baseline and follow-up data registration of patients with a diagnosis of NAFLD/NASH/MAFLD, according to standardized criteria.
  This will allow future studies aimed at elucidate clinical presentation, natural history, response to treatment, genetic and metabolic risk factors, treatment options and outcomes of the disease. The cohort will allow investigators to carry out genetic, serological, microbiologic and immunological studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Epatocentro Ticino, Lugano, Canton Ticino, Switzerland